CLINICAL TRIAL: NCT02902900
Title: Observational Cohort Study Evaluating the Use and Efficacy of Pomalidomide in Patients With Multiple Myeloma in Routine Clinical Practice
Brief Title: An Efficacy Study of Pomalidomide in Patient With Multiple Myeloma in Routine Clinical Practice
Acronym: MIROIR
Status: Completed | Type: Observational
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Other Study IDs: CC-4047-MM-018
Record Dates: First submitted 2016-09-13; First posted 2016-09-16 (Estimated); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Pomalidomide; Efficacy
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Imnovid: Patients relapse/ refractory multiple myeloma who initiated pomalidomide in routine clinical practice

SUMMARY:
This study, a national, multicenter, observational, ambispective, non-interventional study, will be conducted in French hospitals prescribing pomalidomide and already participating in the ongoing Imnovid registry.

This study will add to the registry. Indeed, pomalidomide-prescribing physicians and pharmacists dispensing pomalidomide have to enter into the Imnovid registry all patients who have been prescribed this drug since the date on which it was marketed regardless of the initiation date of pomalidomide or the indication for which it was prescribed.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (age ≥ 18 yrs),
* Diagnosed with multiple myeloma (measurable or not),
* In whom pomalidomide treatment was first initiated between October 1, 2014, and September 30, 2019,
* Patient already included in the Imnovid registry,
* Having received oral and written information about the study, and having given their consent to participate.

Exclusion Criteria:

* Previous participation in a clinical trial with pomalidomide,
* Treatment with pomalidomide in a previous line,
* Simultaneous participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The MIROIR study focuses on multiple myeloma patients treated with pomalidomide in France whose treatment was initiated between October 1, 2014, and September 30, 2019. Patients having initiated pomalidomide outside of this period or having received pomalidomide in a previous treatment line will not be included.
Sampling Method: Non-Probability Sample
Enrollment: 2504 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | Up to approximately 6 months
  Is defined as the time between the date of treatment initiation with pomalidomide and the date of the first progression according to the International Myeloma Working Group (IMWG) criteria or death whatever the cause.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Up to 2 years
  Is defined by at least a partial response (PR) according to IMWG criteria
Duration of Response (DOR) | Up to 2 years
  Is calculated for responders with at least partial response (PR) as the time between the first observation of response and the time of the first event such as disease progression or death due to progression.
Overall Survival (OS) | Up to 2 years
  Is defined as the duration between the date of the start of treatment and the date of death whatever the cause.
Time to Progression (TTP) | Up to 2 years
  Is defined as the time between the start of pomalidomide treatment and disease progression according to IMWG criteria, or death due to progression.
Time to Treatment Failure (TTF) | Up to 2 Years
  Is defined as the duration between the date of the start of pomalidomide treatment and the first progression according to IMWG criteria, second cancer, toxicity requiring treatment discontinuation or death of the patient.
Adverse Events (AEs) | Up to 3 years
  Number of subjects with adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (125):
- France (125):
  - Centre Hospitalier General, Albi
  - Groupe Hospitalier Sud, Amiens
  - Hotel Dieu, Angers
  - Ch D'Arras, Arras
  - Centre Hospitalier Intercommunal Robert Ballanger, Aulnay-sous-Bois
  - Centre Hospitalier H. Duffaut, Avignon
  - Centre Hospitalier Jeanne d'Arc, Bar-le-Duc
  - Chic Cote Basque Bayonne, Bayonne
  - Hopital Nord Franche-Comte - Site de Belfort, Belfort
  - Hopital Jean Minjoz, Besançon
  - Centre Hospitalier General, Blois
  - Hôpital Avicenne, Bobigny
  - Institut Bergonie, Bordeaux
  - Polyclin Bordeaux Nord Aquitaine, Bordeaux
  - Ch Docteur Duchenne, Boulogne-sur-Mer
  - Ch de Fleyriat, Bourg-en-Bresse
  - Ch Pierre Oudot, Bourgoin
  - Hopital Augustin Morvan, Brest
  - Hôpital d'Instruction des Armées, Brest Armees Cedex 9
  - Ch de Brive La Gaillarde, Brive-la-Gaillarde
  - Hopital Cote de Nacre, Caen
  - Hopital Pierre Nouveau, Cannes
  - Clinique Du Parc, Castelnau-le-Lez
  - Hopital Prive Sevigne, Cesson-Sévigné
  - Médipôle de Savoie, Challes-les-Eaux
  - Ch William Morey, Chalon-sur-Saône
  - Ch de Chambery, Chambéry
  - Centre Hospitalier, Cholet
  - Hopital Antoine Beclere, Clamart
  - Chu Estaing, Clermont-Ferrand
  - Pole Sante Republique, Clermont-Ferrand
  - Ch Sud Francilien, Corbeil-Essonnes
  - Centre Hospitalier de Creil, Creil
  - Gh Henri Mondor Albert Chenevier, Créteil
  - Ch de Dax, Dax
  - Hopital Francois Mitterrand, Dijon
  - Ch Dracenie, Draguignan
  - Ch de Dunkerque, Dunkirk
  - Centre Hospitalier Emile Durkheim, Épinal
  - Clinique Pasteur, Évreux
  - Chi de Frejus Saint Raphael, Fréjus
  - Chi Des Alpes Du Sud, Gap
  - Institut Daniel Hollard, Grenoble
  - Hopital Charles Foix, Ivry-sur-Seine
  - Polyclinique de Blois, La Chaussée-Saint-Victor
  - Ch Dptal Les Oudairies, La Roche-sur-Yon
  - Centre Hospitalier de La Rochelle, La Rochelle
  - Hopital Albert Michallon, La Tronche
  - Ch Andre Mignot, Le Chesnay
  - Hopital Louis Pasteur, Le Coudray
  - Clinique Victor Hugo, Le Mans
  - Ch Du Mans, Le Mans
  - Ch Du Docteur Schaffner, Lens
  - Hopital Robert Boulin, Libourne
  - Hopital Saint Vincent, Lille
  - Hopital Claude Huriez, Lille
  - Hopital Dupuytren, Limoges
  - Ch Bretagne Sud Site Lorient, Lorient
  - Centre Hospitalier General, Lourdes
  - Hopital Edouard Herriot, Lyon
  - Institut J Paoli-Calmettes, Marseille
  - Hôpital Saint Joseph, Marseille
  - Hopital de La Conception, Marseille
  - Centre Hospitalier de Martigues, Martigues
  - Ch de Meaux, Meaux
  - Hopital Marc Jacquet, Melun
  - Hopital Belle Isle, Metz
  - HOPITAL Metz Mercy, Metz
  - Hopital Jacques Monod, Montivilliers
  - Clinique Beau Soleil, Montpellier
  - Hopital Saint Eloi, Montpellier
  - Ch Des Pays de Morlaix, Morlaix
  - Ch Mulhouse, Mulhouse
  - Hopital Hotel Dieu Et Hme, Nantes
  - Centre Catherine de Sienne, Nantes
  - Ch Pierre Beregovoy, Nevers
  - Centre Antoine Lacassagne, Nice
  - Hopital de L'Archet, Nice
  - Hopital Caremeau, Nîmes
  - Hopital Saint Louis, Paris
  - Hôpital Saint Antoine, Paris
  - Gh Pitie Salpetriere, Paris
  - Gh Cochin St Vincent de Paul, Paris
  - Hopital Necker Enfants Malades, Paris
  - Hopital Saint Jean, Perpignan
  - Polyclinique Francheville, Périgueux
  - Ch de Perigueux, Périgueux
  - Ch Lyon Sud, Pierre-Bénite
  - Hopital La Miletrie, Poitiers
  - Ch Rene Dubos, Pontoise
  - CH Annecy Genevois, Pringy
  - Chi de Cornouaille, Quimper
  - Ch de Rambouillet, Rambouillet
  - Chu Reims, Reims
  - Hopital Robert Debre, Reims
  - Hopital Pontchaillou, Rennes
  - Chu Rennes - Hopital Sud, Rennes
  - Ch de Roanne, Roanne
  - Hopitaux Drome Nord, Romans-sur-Isère
  - Hopital Victor Provo, Roubaix
  - Centre Henri Becquerel, Rouen
  - Hopital Yves Le Foll, Saint-Brieuc
  - Centre Rene Huguenin, Saint-Cloud
  - Centre Hospitalier General, Saint-Germain-en-Laye
  - Centre Rene Gauducheau, Saint-Herblain
  - Hôpital Nord, Saint-Priest-en-Jarez
  - Institut de Cancérologie de la Loire, Saint-Priest-en-Jarez
  - Chg de Saint Quentin, Saint-Quentin
  - C.H. Jacques Boutard, Saint-Yrieix-la-Perche
  - Centre Hospitalier, Sens
  - Centre Hospitalier, St-Malo
  - Hopital Hautepierre, Strasbourg
  - Hopital Foch, Suresnes
  - C.H.I Les Hopitaux Du Leman, Thonon-les-Bains
  - Hopital Sainte Musse, Toulon
  - Hopital Rangueil, Toulouse
  - IUCT Oncopole, Toulouse
  - Hopital Bretonneau, Tours
  - Hopital Des Hauts Clos, Troyes
  - Centre Hospitalier de Valence, Valence
  - Ch de Valenciennes, Valenciennes
  - Hopitaux de Brabois, Vandœuvre-lès-Nancy
  - Ch Bretagne Atlantique de Vannes, Vannes
  - Chi de La Haute Saone de Vesoul, Vesoul
  - Institut Gustave Roussy, Villejuif

REFERENCES:
- [Background] Waldschmidt JM, Simon A, Wider D, Muller SJ, Follo M, Ihorst G, Decker S, Lorenz J, Chatterjee M, Azab AK, Duyster J, Wasch R, Engelhardt M. CXCL12 and CXCR7 are relevant targets to reverse cell adhesion-mediated drug resistance in multiple myeloma. Br J Haematol. 2017 Oct;179(1):36-49. doi: 10.1111/bjh.14807. Epub 2017 Jul 2. PMID 28670693
- [Background] Dinner S, Dunn TJ, Price E, Coutre SE, Gotlib J, Berube C, Kaufman GP, Medeiros BC, Liedtke M. A phase I, open-label, dose-escalation study of amrubicin in combination with lenalidomide and weekly dexamethasone in previously treated adults with relapsed or refractory multiple myeloma. Int J Hematol. 2018 Sep;108(3):267-273. doi: 10.1007/s12185-018-2468-5. Epub 2018 May 25. PMID 29802551
- [Background] Garderet L, Kuhnowski F, Berge B, Roussel M, Escoffre-Barbe M, Lafon I, Facon T, Leleu X, Karlin L, Perrot A, Moreau P, Marit G, Stoppa AM, Royer B, Chaleteix C, Tiab M, Araujo C, Lenain P, Macro M, Voog E, Benboubker L, Allangba O, Jourdan E, Orsini-Piocelle F, Brechignac S, Eveillard JR, Belhadj K, Wetterwald M, Pegourie B, Jaccard A, Eisenmann JC, Glaisner S, Mohty M, Hulin C, Loiseau HA, Mathiot C, Attal M. Pomalidomide, cyclophosphamide, and dexamethasone for relapsed multiple myeloma. Blood. 2018 Dec 13;132(24):2555-2563. doi: 10.1182/blood-2018-07-863829. Epub 2018 Oct 3. PMID 30282798
- [Background] Mark TM, Forsberg PA, Rossi AC, Pearse RN, Pekle KA, Perry A, Boyer A, Tegnestam L, Jayabalan D, Coleman M, Niesvizky R. Phase 2 study of clarithromycin, pomalidomide, and dexamethasone in relapsed or refractory multiple myeloma. Blood Adv. 2019 Feb 26;3(4):603-611. doi: 10.1182/bloodadvances.2018028027. PMID 30792190
- [Background] Ailawadhi S, DerSarkissian M, Duh MS, Lafeuille MH, Posner G, Ralston S, Zagadailov E, Ba-Mancini A, Rifkin R. Cost Offsets in the Treatment Journeys of Patients With Relapsed/Refractory Multiple Myeloma. Clin Ther. 2019 Mar;41(3):477-493.e7. doi: 10.1016/j.clinthera.2019.01.009. Epub 2019 Feb 14. PMID 30773308
- [Background] Li Y, Wang X, Liu L, Zhang C, Gomez D, Reyes J, Palmisano M, Zhou S. An Open-Label, Phase 1 Study to Assess the Effects of Hepatic Impairment on Pomalidomide Pharmacokinetics. Clin Pharmacol Drug Dev. 2019 Apr;8(3):346-354. doi: 10.1002/cpdd.470. Epub 2018 May 10. PMID 29746728
- See also: Expanded Access for CC-4047 — https://clinicaltrials.gov/ct2/show/NCT03723096?term=NCT03723096&rank=1